CLINICAL TRIAL: NCT07368153
Title: A Randomised, Controlled, Double-blind Study to Evaluate the Safety and Tolerability of IDO-1 Inhibition in the Prevention of EBV-related Pathology in EBV Negative Kidney Transplant Recipients Receiving an Organ From EBV Positive Donors.
Brief Title: Safety and Tolerability of IDO-1 Inhibition in the Prevention of EBV-related Pathology in EBV Negative Kidney Transplant Recipients Receiving an Organ From EBV Positive Donors
Acronym: IDEP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Hornet Therapeutics. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-02366; ub24hess
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: EBV Infections; Kidney Transplant
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: A randomised, controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: indoleamine 2,3-dioxygenase 1 (IDO-1) inhibitor
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: indoleamine 2,3-dioxygenase 1 (IDO-1) inhibitor — Study treatment will be initiated one day prior to kidney transplantation or, for recipients of cadaveric donor organs, on the day of transplantation, and will be administered at a dose of 200 mg once daily for a total duration of 28 days, followed by a safety follow-up phase.
  Arms: Treatment
Drug: placebo — A matching placebo will be administered once daily, initiated one day prior to kidney transplantation or, for recipients of cadaveric donor organs, on the day of transplantation, for a total duration of 28 days, followed by a safety follow-up phase.
  Arms: Placebo

SUMMARY:
This clinical study will evaluate the safety and tolerability of an IDO-1 inhibitor in patients receiving a kidney transplant. The study includes individuals who have not previously been infected with Epstein-Barr virus (EBV) and who receive a kidney from a donor with prior EBV infection.

Participants will receive the IDO-1 inhibitor or placebo in addition to standard medical care and will be monitored for side effects and other safety-related outcomes throughout the study.

DETAILED DESCRIPTION:
This clinical study is being conducted to evaluate the safety and tolerability of an IDO-1 inhibitor in patients receiving a kidney transplant. The study population includes individuals who are Epstein-Barr virus (EBV) seronegative and receive a kidney from an EBV-seropositive donor, a group at increased risk for EBV-related complications following transplantation.

Kidney transplantation requires substantial immunosuppression to maintain graft function. While necessary, this immunosuppression increases susceptibility to infections, including EBV, which may lead to serious clinical consequences in immunocompromised individuals.

In this study, participants will receive the IDO-1 inhibitor or placebo in addition to standard-of-care immunosuppressive therapy. Study treatment will be initiated prior to kidney transplantation or on the day of transplantation, depending on donor availability, and will be administered for a defined treatment period, followed by a safety follow-up phase.

The primary objective of the study is to assess the safety and tolerability of the IDO-1 inhibitor in kidney transplant recipients, including the incidence of adverse events and clinically relevant laboratory abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Male or female aged ≥18 years
3. EBV seronegative at the time of renal transplant
4. If women of child-bearing potential (WOCBP), participants must have a negative serum pregnancy test at screening and inclusion, and must be willing to use a highly effective method of birth control for the duration of the study. Acceptable methods of contraception:

   1. Hormonal contraception associated with inhibition of ovulation
   2. Intrauterine device (IUD)
   3. Intrauterine hormone-releasing system (IUS)
   4. Bilateral tubal occlusion
   5. Vasectomised partner
   6. Condom with spermicide
   7. Sexual abstinence, in line with the preferred and usual lifestyle of the participant. Periodic abstinence (such as calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
5. If male, participants must be prepared to use reliable barrier method contraception and a second method such as spermicide for the duration of the study unless surgically sterile.

Exclusion Criteria:

1. EBV seropositivity at the time of transplant
2. Participants with any form of cancer within the last 12 months, or patients continuing to receive chemo or immunotherapy within the last 12 months.
3. Participants with a history of PTLD
4. Other active systemic infections requiring treatment prior to and at the time of baseline. Prophylactic agents are permitted.
5. CYP3A4 and CYP2C28 Inhibitors and Inducers (List may be found in Appendix 1)
6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥3 x ULN
7. Any condition for which, in the opinion of the investigator, the treatment or participation in the study may pose a health risk to the participant
8. Planned or active participation in any other study with an investigational medicinal product (IMP).
9. Have taken an IMP within the last 3 months.
10. Unwilling or unable to provide fully informed consent.
11. Unwilling or unable to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 12 weeks post-treatment
Incidence of serious adverse events | up to 12 weeks post-treatment
Number of participants experiencing adverse events | up to 12 weeks post-treatment
Number of participants experiencing clinically significant changes in safety assessments | up to 12 weeks post-treatment
  Safety assessments include vital signs (pulse rate, blood pressure, and body temperature), 12-lead electrocardiogram (ECG), and laboratory evaluations (haematology and serum/plasma biochemistry), assessed up to and including 12 weeks post-treatment.

SECONDARY OUTCOMES:
Changes in EBV viral load | up to 12 weeks post-treatment
  Assessment EBV viral load in the event of a primary EBV infection
Changes in EBV viral dynamics | up to 12 weeks post-treatment
  Assessment of EBV viral dynamics in the event of a primary EBV infection
Exploratory metabolomic analysis | up to 12 weeks post-treatment
  including parameters related to the kynurenine pathway
Exploratory analysis peripheral blood mononuclear cells (PBMCs) | up to 12 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Diebold, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No